CLINICAL TRIAL: NCT00206063
Title: Long-Term Treatment With the Oral Direct Thrombin Inhibitor Ximelagatran, Compared to Warfarin, as Stroke Prophylaxis in Patients With Atrial Fibrillation. A Long Term Follow-Up Study
Brief Title: Long Term Open Follow-up With H376/95 vs. Warfarin
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Melagatran/ximelagatran was withdrawn from the market and clinical development in February 2006 in the interest of patient safety.
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SH-TPA-0004; D4004C00004
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2010-11-15 (Estimated); Status verified 2010-11

CONDITIONS: Stroke Prevention in Patients With Atrial Fibrillation
MeSH Terms: interventions — ximelagatran

INTERVENTIONS:
Drug: EXANTA
  Other Names: Ximelagatran

SUMMARY:
The purpose of this study is to evaluate tolerability of long-term treatment with ximelagatran compared to standard treatment with warfarin.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Completion of the study SH-TPA-0002, history of chronic atrial fibrillation (i.e. rapidly beating heart), at least one risk factor for stroke (e.g. high blood pressure, age over 65, previous stroke or similar attack, diabetes or coronary heart disease)

Exclusion Criteria:

* Conditions associated with increased risk of bleeding, renal impairment, known active liver disease or liver insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220
Dates: Start 1999-08; Primary Completion 2004-06 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events, with special regard to bleeding, thromboembolic events and discontinuation of treatment.

CONTACTS AND LOCATIONS:
Locations (19):
- Research Site, Palo Alto, California, United States
- Research Site, Oostduinkerke, Belgium
- Czechia (5):
  - Research Site, Helsingor
  - Research Site, Most
  - Research Site, Plzeo
  - Research Site, Poibram
  - Research Site, Prague
- Denmark (2):
  - Research Site, Aarhus
  - Research Site, Odense
- Finland (2):
  - Research Site, Kuopio
  - Research Site, Savonlinna
- Norway (2):
  - Research Site, Hamar
  - Research Site, Oslo
- Poland (3):
  - Research Site, Płock
  - Research Site, Siedice
  - Research Site, Warsaw
- Research Site, Lund, Sweden
- United Kingdom (2):
  - Research Site, Leicester
  - Research Site, Newcastle